CLINICAL TRIAL: NCT03685409
Title: Cancer Chemoprevention by Metformin Hydrochloride Compared to Placebo in Oral Potentially Malignant Lesions: A Randomized Clinical Trial (Part 1)
Brief Title: Cancer Chemoprevention by Metformin Hydrochloride in Oral Potentially Malignant Lesions
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Mohamed Abdelazim, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 023836530
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin-Group (Active Comparator): Metformin hydrochloride tablets 500 mg taken orally once daily for 3 months
  Interventions: Drug: Metformin Hydrochloride 500 MG
- Placebo-Group (Placebo Comparator): Starch placebo tablets taken orally once daily for 3 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metformin Hydrochloride 500 MG — Metformin hydrochloride tablets 500 mg given orally once daily.
  Other Names: Glucophage; Cidophage
  Arms: Metformin-Group
Drug: Placebo Oral Tablet — Starch Placebo oral tablets will be given once daily to the control group
  Arms: Placebo-Group

SUMMARY:
Oral squamous cell carcinomas (OSCCs) are among the most common types of head and neck cancers and are a major cause of significant morbidity. It was reported that 16- 62% of OSCCs develop from premalignant lesions, which often presents clinically as white or red mucosal patches known as leukoplakia and erythroplakia.

The role of miRNA in cancer has been established by many studies that have shown that miRNA signatures (i.e., mRNA expression profiles) can be useful for classifying human cancers. These studies have identified "cancer related miRNAs through investigating expression profiles in matched normal and tumor tissues, as well as in body fluids.

Metformin, one of most widely prescribed oral hypoglycemic agents, has recently received increased attention because of its potential anti-tumorigenic effects that are thought to be independent of its hypoglycemic effects. Evans et al. first found an association between metformin use and decreased cancer incidence.

The study will reveal whether Systemic Metformin hydrochloride treatment given to patients with oral potentially malignant lesions improve the prognosis and prevent or at least reduce the incidence of malignant transformation?

DETAILED DESCRIPTION:
The idea of identifying oral lesions with a precancerous nature, that is, in the sense of pertaining to a pathologic process with an increased risk for future malignant development, of course, is to prevent frank malignancy to occur in the affected area.

In 2005, WHO categorized any lesion or condition that may increase the risk of malignant transformation as an 'oral potentially malignant disorder' (OPMD). Early detection of cancer development from oral premalignant lesions (OPLs) plays an important role in successful therapy. The management of OPMDs varies according to the type of lesion and often differs between treatment centers. However, it remains unclear if excision of leukoplakia/erythroplakia protects patients against the development of OSCC and no randomized controlled trials have been performed to address this issue.

Various treatment modalities, such as systemic therapies and surgical removal, have been suggested. The systemic therapies tested so far include retinoids, extracts of green tea, inhibitors of cyclooxygenase-2 and of epidermal growth factor, and peroxisome proliferator-activated receptor-c agonists, but there is no generally approved standard systemic therapy regimen so far.

Local removal includes photodynamic therapy, laser therapy, cryotherapy and conventional removal by scalpel, but no treatment has so far gained universal approval, no treatment has so far been subjected to a randomized clinical trial (RCT), and no treatment has been shown to prevent recurrence or significantly reduce malignant development in long-term follow-up studies. It is well established that no treatment results in malignant development at an annual rate of 2-3%.

The overall purpose of treatment therefore is to reduce this percentage. However, the situation is to take responsibility for the welfare of the patients still is, as it has been so far: despite treatment, in some types of lesions cancers do occur, so the important question is whether the harm to patients by not treating or by treating them? Lack of randomized clinical trials accounts for this persistent question, and while waiting for such studies to be reported, it is necessary to reflect on the existing scenarios.

Field cancerization To explain why surgery may not always be beneficial, it has been mentioned that the visible lesions may be surrounded by genetically altered, cancer stigmatized epithelial cells unrevealed by routine clinical inspection and histological examination. A possible outcome of such characteristics is obviously lacking resection of all affected tissue with recurrence and development of carcinoma from residual genetically altered cells.

Introduction to MicroRNA MicroRNAs (miRNAs) are non-coding regulatory RNA molecules of 19-25 nucleotides in length. miRNAs play a major role in maintaining tissue homeostasis by regulating many processes such as cellular proliferation, differentiation, migration, apoptosis, survival and morphogenesis.

It is estimated that the human genome may harbor up to 1,000 miRNAs. Although miRNAs are not directly involved in encoding proteins, they are believed to control the expression of more than one third of all protein coding genes present within the human genome. Historically, miRNAs have been viewed as negative regulators of gene expression. Recent work by Vasudevan et al., has, however, shown that a small subset of miRNAs within the human genome can also enhance gene expression.

Role of miRNAs in cancer The role of miRNA in cancer has been reiterated and established by many studies that have shown that miRNA signatures (i.e., mRNA expression profiles) can be useful for classifying human cancers. These studies have identified "cancer related miRNAs" through investigating expression profiles in matched normal and tumor tissues, as well as in body fluids. In addition, a vast number of studies have shown that miRNAs can play a role in regulating the expression of oncogenes and tumor suppressor genes, whereas others have shown that miRNA gene deletion or mutation can lead cancer initiation, progression and metastasis. Calin et al., were the first to demonstrate that a differential expression of miRNAs may provide useful tools in the diagnosis and prognosis of human cancers.

MicroRNAs as diagnostic tools Many miRNAs are uniquely and differentially expressed in certain tissues as compared with normal adjacent tissues. These small RNA molecules can have diagnostic or prognostic value, as miRNA expression profiles reflect tumor origin, stage, and other pathological factors. For example, the expression of miRNA let-7 is downregulated in lung cancer but not in other cancers, such as breast or colon cancer. These observations suggest that miRNAs can be used as biomarkers and diagnostic tools for cancer detection. Moreover, miRNAs can function as accurate molecular markers also because they are relatively stable and resistant to RNase degradation-probably due to their small size.

miR-21 and miR-200 seem to be particularly relevant to OSCC. Inhibition of miR-21 in tongue cancer cells in vitro reduces survival and anchorage-independent growth. miR-21 increases proliferation, migration and anchorage-independent growth of HNSCC cells in vitro and in mouse models, thereby augmenting the oncogenic potential of these cells.

Detection of miRNAs in body fluids With the advances of molecular biological techniques and the increasing knowledge of tumor pathogenesis, bio-markers are now considered as an effective supplement, in conjunction to histological examination, for facilitating clinical decision making. Extracellular miRNAs in serum, plasma, saliva and urine have recently been shown to be associated with various pathological conditions, including cancer. Most of the circulating miRNAs are included in lipid or lipoprotein complexes, such as apoptotic bodies, micro vesicles or exosomes, rendering them inaccessible to degradation by RNAses. Lawrie and colleagues were the first to observe elevated levels of miRNA-21 in serum samples collected from large B-cell lymphoma patients.

Explanation for choice of comparators:

Control/comparator : Patients receiving the standard of care together with PLACEBO starch tablets.

Management strategies for patients with OPLs fall into three categories: close observation, surgical removal and ablation, and medical therapies. The mainstay of therapy is observation using frequent clinical examinations. The frequency of examinations should be tailored to individual patient factors such as the clinical appearance and stage of lesion; presence of dysplasia; continued use of tobacco, alcohol, or Areca quid; reliability; and access to medical care.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with age range from 20 to 70 years.
* Patients able to return for the follow up visits and can perform oral hygiene measures.
* Clinically diagnosed and histologically confirmed as having oral potentially malignant lesions (Atrophic oral lichen planus, leukoplakia, erythroplakia and oral submucous fibrosis).
* Patients agreed to sign a written consent after understanding the nature of the study
* Patients have diagnosed oral premalignant lesion/lesions and not yet turned into malignancy

Exclusion Criteria:

* Diabetic patients (Diabetes Mellitus Type I & II)
* Patients have cardiovascular, lung, Renal, Liver diseases
* Patients on H2 blocker & proton pump inhibitors therapy as Ranitidine (affects metformin absorption and clearance)
* Those with allergy or sensitivity to Metformin therapy or having any contraindication for their use.
* Systemic and/or local systemic drug therapy within the last 3 months prior to the start of the study
* Patients on steroidal or Non-steroidal anti-inflammatory drugs (NSAIDs) for at least the last 6 months
* Patients on Antibiotics treatment for at least the last 2 months
* Patients on Retinoid, green tea supplements or another natural products therapy
* Patients with already diagnosed malignant lesion/lesions
* Pregnant or Lactating females
* Vulnerable groups as prisoners, mentally disabled, etc…

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes | 3 months
  Effect of Systemic Metformin hydrochloride on the millimeters change in the largest diameter of the oral potentially malignant lesion

SECONDARY OUTCOMES:
Immunohistochemical analysis | 3 months
  Numerical change in immunohistochemical expression of Cyclin-D1 at baseline and at 3 months after using Metformin using computer aided image analysis
microRNA analysis | 3 months
  Numerical differences between miR-21 and miR-200 at baseline and at 3 months using Realtime PCR
Salivary microRNA | 3 months
  Numerical difference between the expression of miR-21 and miR-200 in tissue biopsies Versus Saliva at baseline and at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided